CLINICAL TRIAL: NCT07384546
Title: Spontaneous Breathing-Preserved Anesthesia and Surgical Strategy to Improve Early Postoperative Hospital Recovery After Lung Transplantation (BREATHE), A Prospective, Multicenter, Blinded Endpoint Assessment Single-arm Clinical Study
Brief Title: BREATHE Study: Spontaneous Breathing-Preserved Anesthesia and Surgical Strategy for Hospital Recovery in Lung Transplantation
Acronym: BREATHE-LTx
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Chief Physician and Professor of Thoracic Surgery, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BREATHE-LTx-Study
Record Dates: First submitted 2025-12-01; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: End-stage Lung Disease
Keywords: Lung transplantation; Enhanced Recovery After Surgery

STUDY DESIGN:
Masking Description: Outcome assessors (and statisticians, if applicable) will be blinded to intraoperative airway management and ventilation details.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tubeless LTx Group (Experimental): Single-group arm. All participants receive lung transplantation under a standardized spontaneous-breathing-preserving ("tubeless") pathway. After anesthesia induction, a supraglottic airway (laryngeal mask airway) is used when feasible with regional nerve blocks and multimodal sedation/analgesia to control pain and cough while maintaining spontaneous breathing. Muscle relaxants are minimized; ventilatory assistance is provided only as needed with low airway pressures. Postoperatively, patients are managed in the intensive care unit with spontaneous breathing and protocol-guided noninvasive respiratory support. Conversion to endotracheal intubation, invasive mechanical ventilation, and/or extracorporeal membrane oxygenation is allowed if predefined safety criteria are met.
  Interventions: Procedure: Lung transplantation that preserves spontaneous breathing function

INTERVENTIONS:
Procedure: Lung transplantation that preserves spontaneous breathing function — This intervention uses a spontaneous-breathing-preserving anesthesia strategy during lung transplantation, which differs from conventional management based on endotracheal intubation and invasive mechanical ventilation.
  A supraglottic airway (laryngeal mask airway) is used when feasible instead of endotracheal intubation to maintain spontaneous breathing throughout the procedure.
  Neuromuscular blocking agents are minimized, and regional nerve blocks (such as intercostal nerve blocks or paravertebral blocks) are used to control pain and suppress cough while preserving the patient's ability to breathe independently.
  After surgery, patients receive protocol-guided noninvasive respiratory support (for example, high-flow nasal oxygen or noninvasive ventilation), with the goal of avoiding routine invasive mechanical ventilation.

SUMMARY:
The goal of this study is to learn whether a spontaneous-breathing ("tubeless") anesthesia and surgery strategy can improve early recovery and remain safe for adults who receive a lung transplant. This strategy aims to help lung transplant recipients maintain spontaneous breathing as much as possible during and after surgery, avoid tracheal intubation with invasive mechanical ventilation and deep sedation, and thereby support faster recovery while maintaining postoperative survival and safety. All participants will receive lung transplantation supported by the same spontaneous-breathing ("tubeless") strategy. Researchers plan to enroll about 110 participants at several hospitals in China. A separate study team will review the main outcomes using predefined study rules.

The main questions this study aims to answer are: The main questions this study aims to answer are: among adult lung transplant recipients, does an anesthesia-surgical strategy that preserves spontaneous breathing improve early postoperative recovery while remaining safe during the first 30 days after surgery? The study will focus on the need for postoperative invasive mechanical ventilation, length of postoperative hospital stays, and in-hospital mortality.

Participants will: Complete screening tests and assessments before surgery (up to about 30 days before the transplant). Undergo lung transplantation using a standardized approach that aims to keep spontaneous breathing function, often using a laryngeal mask airway instead of a breathing tube. Receive pain and cough control measures (such as local anesthesia or nerve block anesthesia) and close monitoring during and after surgery. Receive standard postoperative care. If safety concerns arise, the clinical team will use invasive mechanical ventilation or extracorporeal membrane oxygenation when needed. Be followed during the hospital stay and for 90 days after surgery to record recovery, complications, and readmissions.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm clinical study designed to evaluate a standardized perioperative pathway for adult lung transplantation that aims to preserve spontaneous breathing ("tubeless" strategy). The study will enroll approximately 110 participants across multiple hospitals in China. To reduce assessment bias in a single-arm design, key study endpoints will be evaluated by an independent team using prespecified definitions and adjudication rules.

The investigational perioperative pathway integrates anesthesia and surgical management with the goal of maintaining the participant's own breathing as much as possible during and after transplantation, while minimizing exposure to tracheal intubation, invasive mechanical ventilation (IMV), and deep sedation. The approach typically uses a laryngeal mask airway (LMA) for airway support, intravenous anesthesia with careful titration, and multimodal analgesia to achieve adequate comfort and cough control while allowing spontaneous respiration. Regional and/or local anesthetic techniques may be used to improve pain control and reduce airway stimulation. Intraoperative monitoring and ventilatory support are individualized, and lung recruitment or short periods of assisted ventilation may be used when clinically indicated.

Participant safety is prioritized throughout the procedure and postoperative period. The clinical team may convert to conventional tracheal intubation and IMV at any time if predefined clinical concerns arise, such as inadequate gas exchange, airway protection issues, hemodynamic instability, uncontrolled bleeding, or conditions that compromise surgical safety. Extracorporeal membrane oxygenation (ECMO) may be initiated or escalated when necessary according to institutional practice and prespecified clinical triggers. Postoperatively, participants receive standard transplant care per each center's routine protocols, including intensive monitoring and timely escalation of respiratory or circulatory support when required.

The study timeline includes a screening period prior to transplantation, comprehensive perioperative data capture, in-hospital follow-up through discharge, and structured follow-up after discharge to document early recovery and safety outcomes. Safety surveillance focuses on events occurring within 30 days after transplantation, and additional follow-up through 90 days captures short-term outcomes such as survival status and rehospitalization.

All study data are recorded in standardized case report forms and entered into a centralized database with built-in quality checks. The coordinating center oversees data completeness and consistency across sites, and the independent outcome review team adjudicates endpoints according to prespecified rules.

ELIGIBILITY:
【1】Inclusion Criteria

1. Age and informed consent: Aged 18-70 years; able to understand the study and provide written informed consent; willing and able to complete follow-up.
2. Transplant candidacy: Listed in the CLuTR registry and/or the local center's lung transplant waiting list, and scheduled to undergo allogeneic lung transplantation.
3. Preoperative support status: Not on ongoing invasive mechanical ventilation preoperatively (endotracheal intubation or tracheostomy), and not receiving ECMO or other extracorporeal life support.
4. Minimum key organ function requirements: LVEF ≥40%; eGFR ≥40 mL/min/1.73 m²; no acute liver failure and no evidence of decompensated cirrhosis/portal hypertension; ASA Physical Status (American Society of Anesthesiologists classification) ≤ IV.
5. Infection and transmissible diseases: No evidence of active infection; no active tuberculosis; HIV/HBV/HCV status meeting the center's transplant requirements (e.g., undetectable viral load, noticeability per center policy).
6. Rehabilitation potential and support: Demonstrates postoperative rehabilitation potential (able to cooperate with training) and has reliable caregiving support (at least one primary caregiver).

【2】Exclusion Criteria

1. Informed consent/adherence: Refusal of or withdrawal of informed consent; investigator judgment that the participant cannot complete follow-up or has recurrent severe non-adherence.
2. Transplant type: Re-transplantation, multi-organ transplantation, or planned lobar lung transplantation.
3. Recent major cardiovascular/cerebrovascular events: Acute coronary syndrome/myocardial infarction or stroke within the past 30 days.
4. Severe organ dysfunction/acute failure: LVEF <40%; eGFR <40 mL/min/1.73 m²; acute liver failure or decompensated cirrhosis/portal hypertension; acute kidney failure requiring dialysis with low likelihood of recovery; significant preoperative neuropsychiatric disorders or altered consciousness.
5. High risk of severe infection: Septic shock; active extrapulmonary or disseminated infection; active tuberculosis; detectable HIV viral load (or otherwise not meeting the center's transplant criteria).
6. High bleeding risk: Severe bronchiectasis in which preoperative vascular intervention has not been performed or bleeding risk cannot be adequately mitigated.
7. Malignancy: Active malignancy or malignancy associated with a high risk of recurrence or cancer-related mortality.
8. Extreme body habitus: BMI ≥35 kg/m² or BMI <16 kg/m²; or a confirmed diagnosis of severe chest wall deformity or spinal deformity.
9. Substance use/dependence: Current use of cigarettes, e-cigarettes/vaping, smoked cannabis, or intravenous drug use.
10. Tubeless/spontaneous-breathing strategy not safely feasible: The anesthesia team determines that a difficult airway is anticipated or that laryngeal mask airway (LMA)/non-intubated airway management is unsafe (e.g., expected intraoperative airway difficulty, pharyngeal/laryngeal stenosis unsuitable for LMA), including but not limited to: Mallampati class >III, mouth opening <3 cm, thyromental distance <5 cm, or significant airway anatomical variation (e.g., anomalous right upper lobe bronchial takeoff in candidates for right lung transplantation) deemed difficult to manage safely with an LMA or single-lumen airway.
11. Donor/donor-lung limitations: Donor age >60 years; donor mechanical ventilation >14 days; positive donor-lung airway culture deemed unacceptable by the transplant team.
12. Protected populations: Pregnant or breastfeeding women.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Requiring Postoperative Invasive Mechanical Ventilation (IMV) During Index Hospitalization | From ICU admission immediately after leaving the operating room until hospital discharge or in-hospital death, assessed up to 90 days postoperatively (if hospitalization extends beyond 90 days, events after day 90 will not be counted for this outcome).
  Number of participants who require postoperative invasive mechanical ventilation (IMV) delivered via an endotracheal tube or tracheostomy tube at any time after leaving the operating room and before hospital discharge (including in-hospital death).
Postoperative Hospital Length of Stay (Days) During Index Hospitalization | From end of surgery (postoperative Day 0) until hospital discharge or in-hospital death (index hospitalization), assessed up to 90 days.
  the number of days from the end of surgery (postoperative Day 0) to the date the participant is discharged from the index hospitalization, according to institutional discharge criteria. Participants who die in hospital will be assigned length of stay through the date of in-hospital death.
Rate of Perioperative Survival | From start of transplant surgery through hospital discharge or postoperative Day 30, whichever occurs first.
  Perioperative survival is defined as the proportion of participants who remain alive from the start of transplant surgery through hospital discharge or postoperative Day 30, whichever occurs first. Participants who die before discharge or before postoperative Day 30 will be counted as non-survivors for this outcome.

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual participant data (IPD) underlying the analyses of this clinical study, limited to baseline and perioperative variables. Baseline IPD will include demographics (e.g., age, sex), primary diagnosis, key comorbidities, and transplant-relevant preoperative measures and donor/recipient characteristics recorded in structured fields. Perioperative IPD will include operative and anesthesia strategy, airway management, intraoperative/early postoperative respiratory and hemodynamic parameters, major perioperative interventions (e.g., ECMO use), and key in-hospital outcomes during the index hospitalization (e.g., need for postoperative IMV, complications, ICU/hospital length of stay, and in-hospital mortality). The study protocol and statistical analysis plan will also be shared. All direct identifiers will be removed and dates will be shifted/aggregated as needed to protect privacy.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning at study completion and ending 2 years after study completion.
Access Criteria: De-identified IPD and supporting documents (study protocol, statistical analysis plan, and data dictionary) will be available to qualified researchers outside the primary study group for scientifically sound research purposes. Access will be granted upon submission of a written request that includes a brief research proposal, analysis plan, and proof of relevant ethics/IRB review if applicable. Requests will be reviewed by the study steering committee/data access committee. Approved requestors must sign a data use agreement prohibiting re-identification attempts and onward sharing, and requiring appropriate data security measures and acknowledgement of the original study. Data will be provided through a secure electronic transfer or a controlled-access online repository; access instructions will be provided after approval.
URL: https://www.gyfyyy.cn/